CLINICAL TRIAL: NCT05699486
Title: An Open-Label, Multicenter Study To Evaluate the Dose, Efficacy, Safety and Tolerability of PDNO (Nitrosooxypropanol) Infusion in Patients With Pulmonary Hypertension After Cardiopulmonary Bypass (CPB) Surgery for Coronary Artery Bypass Grafting (CABG) or Mitral or Aortic Valve Repair or Replacement With or Without CABG
Brief Title: A Study to Evaluate the Efficacy, Safety and Tolerability of PDNO Infusion in Patients With Pulmonary Hypertension After Cardiopulmonary Bypass Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Attgeno AB (Industry)
Collaborators: Aurevia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-PDNO-003; 2021-005032-30 (EudraCT Number)
Record Dates: First submitted 2022-12-19; First posted 2023-01-26 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Pulmonary Hypertension
Keywords: Acute pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — 1-(nitrosooxy)propan-2-ol and 2-(nitrosooxy)propan-1-ol drug combination; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with PDNO (placebo during baseline and washout observation periods before & after PDNO) (Experimental): PDNO will be administered as an incremental intravenous infusion of respectively 15 minutes with the planned dosage: 3, 10, 30, 45 and 60 nmol/kg/min. If no effect on MPAP/PVR is seen at 60 nmol/kg/min in the first patients treated, further dose escalation up to 120 nmol/kg/min is possible, if recommended by the Internal Safety Review Committe (iSRC) following careful review of collected safety data. The iSRC will in any case review all collected data after 4, 8 and 12 patients (if applicable also after 16 and 20 patients). PDNO is administered together with a carrier buffer (NaHCO3-) flow into a central venous catheter. Placebo (NaCl, commercially available dilution solution for parenteral use, 9 mg/mL) will be administered during the baseline and washout observation periods before and after start of IMP infusion.
  Interventions: Drug: PDNO; Drug: Sodium chloride (placebo)

INTERVENTIONS:
Drug: PDNO — PDNO consists of propylene glycol (1,2-propanediol, PD) chemically combined with NO (to be donated). The drug substance is formulated as an inherent mixture of 4 structure analogues. The mixture consists of an equilibrium of the 2 regioisomers 1-(nitrosooxy) propan-2-ol and 2-(nitrosooxy) propan-1-ol. In addition, each regioisomer is a racemic mixture.
  Other Names: Nitrosooxypropanol
Drug: Sodium chloride (placebo) — Placebo (NaCl, commercially available dilution solution for parenteral use, 9 mg/mL)
  Other Names: NaCl

SUMMARY:
This is an open-label, multicenter study evaluating the dose, effect, safety and tolerability of intravenous PDNO infusion given to patients undergoing cardiopulmonary bypass (CPB) surgery with post-operative acute pulmonary hypertension (aPH).

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willing to sign an informed consent form (ICF)
* Male and female patients, age ≥ 18 years
* Planned to undergo elective cardiopulmonary bypass (CPB) for coronary artery bypass grafting (CABG), aortic valve repair (AVR) or mitral valve repair (MVR) with or without CABG
* Diagnosed with echocardiographic signs of pulmonary artery systolic pressure (PASP) >50 mmHg , as estimated by doppler defined echocardiography using a modified Bernoulli equation: PASP ≈ 4 (tricuspid regurgitant jet velocity)^2 + central venous pressure (CVP)

Exclusion Criteria:

* History of chronic pulmonary hypertension (PH) (WHO group 1, 3, 4 or 5), not group 2 due to left heart disease
* Patients with contraindications for pulmonary artery catheter (PAC)
* History of severe chronic obstructive pulmonary disease
* Left heart failure with ejection fraction (EF) <35%
* Non-ST elevation myocardial infarction (non-STEMI) or ST elevation myocardial infarction (STEMI) within 1 months prior to informed consent
* Stroke (cerebrovascular lesion [CVL]), transient ischemic attack (TIA), AV block III within 3 months prior to informed consent or QTcF >450ms at the time of screening
* High inotropic requirement (no more than one inotrope treatment and the vasopressor norepinephrine at time of screening/postoperative evaluation)
* (Increased) mediastinal bleeding >100 mL/hour in mediastinal drainage at postoperative evaluation
* Mechanical circulatory assistance (intra aortic balloon pump [IABP] or right/left-ventricular assist device [R/L VAD])
* Echocardiographic evidence of significant tricuspid insufficiency
* Body Mass Index (BMI) >40 kg/m^2
* Estimated glomerular filtration rate (eGFR) < 30 mL/min preoperative value
* Methemoglobin >3%
* Indication of liver disease, defined by serum levels of either alanine aminotransferase (ALT), aspartate aminotransferase (AST) or alkaline phosphatase (ALP) above 3 x upper limit of normal (ULN) (preoperative value)
* Preoperative haemoglobin <10 g/dL, postoperative: Hb < 9 g/dL
* Thrombocytopenia (platelet count <100,000/mm^3), preoperative value
* Prothrombin time International ratio (INR) > 1.3, preoperative value
* Pregnant or lactating women, or with a positive pregnancy test at screening (for fertile women only)
* Ongoing daily treatment the last 3 days with non-steroidal anti-inflammatory drugs (NSAIDs, excluding low dose, i.e. 75 mg, acetylsalicylic acid), new oral anticoagulants (NOACs), warfarin, heparin, clopidogrel (last 5 days). Low molecular weight heparin (LMWH) is not an exclusion criterion. Any use of PDE5 inhibitors (sildenafil, tadalafil, vardenafil and avanafil) within 48 hours prior to the administration of PDNO.
* Known active malignancy within the past 3 years except for localized prostate cancer, cervical carcinoma in situ, breast cancer in situ, or nonmelanoma skin cancer that has been definitively treated
* History of allergy/hypersensitivity to PD or ongoing allergy/hypersensitivity or history of hypersensitivity to drugs with a similar chemical structure or class to PDNO
* History of any other clinically significant disease or disorder
* Participation in any interventional clinical study or has been treated with any investigational research products within 30 days or 5 half-lives, whichever is longer, prior to the initiation of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-10-23 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in pulmonary vascular resistance (PVR) | From baseline (mean of -15 minutes and 0 minutes) to time point 15, 30, 45, 60, and 75 minutes with PDNO, respectively; and 85 and 95 minutes with placebo.
  PVR, will be derived as the mean pulmonary artery pressure (MPAP) - pulmonary capillary wedge pressure (PCWP) divided by cardiac output (CO), (PVR=(MPAP-PCWP)/CO), as measured with a pulmonary artery catheter (PAC) including thermodilution-determined cardiac output. Assessments will be done at the following timepoints: T0 (-15 minutes) and T1 (0 minutes) with placebo; T2 (15 minutes), T3 (30 minutes), T4 (45 minutes), T5 (60 minutes), and T6 (75 minutes) with 3, 10, 30, 45, 60 nmol/kg/min with PDNO, respectively; and T7 (85 minutes) and T8 (95 minutes) with placebo.

SECONDARY OUTCOMES:
Mean change in the pulmonary vascular resistance/systemic vascular resistance ratio (PVR/SVR ratio) | From baseline (mean of -15 minutes and 0 minutes) to time point 15, 30, 45, 60, and 75 minutes with PDNO, respectively; and 85 and 95 minutes with placebo.
  PVR, will be derived as the mean pulmonary artery pressure (MPAP) - pulmonary capillary wedge pressure (PCWP) divided by cardiac output (CO), (PVR=(MPAP-PCWP)/CO), as measured with a pulmonary artery catheter (PAC) including thermodilution-determined cardiac output.
  SVR is determined from mean pulmonary artery pressure - central venous pressure divided by cardiac output (CO), (SVR=(MABP-CVP)/CO).
  Assessments will be done at the following timepoints: T0 (-15 minutes) and T1 (0 minutes) with placebo; T2 (15 minutes), T3 (30 minutes), T4 (45 minutes), T5 (60 minutes), and T6 (75 minutes) with 3, 10, 30, 45, 60 nmol/kg/min with PDNO, respectively; and T7 (85 minutes) and T8 (95 minutes) with placebo.
Mean change in fractional area change (FAC) | From baseline (mean of -15 minutes and 0 minutes) to time point 15, 30, 45, 60, and 75 minutes with PDNO, respectively; and 85 and 95 minutes with placebo.
  Assessments will be done at the following timepoints: T0 (-15 minutes) and T1 (0 minutes) with placebo; T2 (15 minutes), T3 (30 minutes), T4 (45 minutes), T5 (60 minutes), and T6 (75 minutes) with 3, 10, 30, 45, 60 nmol/kg/min with PDNO, respectively; and T7 (85 minutes) and T8 (95 minutes) with placebo.
Mean change in tricuspidannular plane systolic excursion (TAPSE) | From baseline (mean of -15 minutes and 0 minutes) to time point 15, 30, 45, 60, and 75 minutes with PDNO, respectively; and 85 and 95 minutes with placebo.
  Assessments will be done at the following timepoints: T0 (-15 minutes) and T1 (0 minutes) with placebo; T2 (15 minutes), T3 (30 minutes), T4 (45 minutes), T5 (60 minutes), and T6 (75 minutes) with 3, 10, 30, 45, 60 nmol/kg/min with PDNO, respectively; and T7 (85 minutes) and T8 (95 minutes) with placebo.
Mean change in right ventricular (RV) free wall strain | From baseline (mean of -15 minutes and 0 minutes) to time point 15, 30, 45, 60, and 75 minutes with PDNO, respectively; and 85 and 95 minutes with placebo.
  Assessments will be done at the following timepoints: T0 (-15 minutes) and T1 (0 minutes) with placebo; T2 (15 minutes), T3 (30 minutes), T4 (45 minutes), T5 (60 minutes), and T6 (75 minutes) with 3, 10, 30, 45, 60 nmol/kg/min with PDNO, respectively; and T7 (85 minutes) and T8 (95 minutes) with placebo.
Safety and tolerability of PDNO in patients undergoing Cardiopulmonary Bypass (CPB) surgery | Until study end (i.e., end of Day 1 [95 minutes]). All AEs (including SAEs) will be collected from the initiation of any study specific procedure, starting when postoperative preparatory preparations are performed on Day 1 and until the end of the study.
  Measured by incidence of: treatment-emergent adverse events (AEs), treatment-emergent serious AEs (SAEs), treatment-emergent AEs of special interest (AESI), treatment-emergent changes in vital signs (blood pressure, pulse, oxygen saturation, respiratory frequency, body temperature), treatment-emergent electrocardiogram (ECG) abnormalities, and treatment-emergent laboratory abnormalities.
Exposure parameters for 1,2-propanediol (PD): estimated area under the curve from time 0 to time t (AUC0-t) | Assessments at time points T0 (-15 minutes; placebo), T6 (75 minutes; PDNO), and T8 (95 minutes; placebo).
  To assess the exposure of PD.
Exposure parameters for 1,2-propanediol (PD): estimated area under the curve from time 0 to infinity (AUC0-inf) | Assessments at time points T0 (-15 minutes; placebo), T6 (75 minutes; PDNO), and T8 (95 minutes; placebo).
  To assess the exposure of PD.
Exposure parameters for 1,2-propanediol (PD): maximum plasma concentration (Cmax) | Assessments at time points T0 (-15 minutes; placebo), T6 (75 minutes; PDNO), and T8 (95 minutes; placebo).
  To assess the exposure of PD.
Exposure parameters for 1,2-propanediol (PD): estimated elimination half life (t½) | Assessments at time points T0 (-15 minutes; placebo), T6 (75 minutes; PDNO), and T8 (95 minutes; placebo).
  To assess the exposure of PD.

OTHER OUTCOMES:
Assess the levels of the following biomarkers: nitrite and nitrate in plasma (µM) | Change from baseline T0 (-15 minutes; placebo) to time point T6 (75 minutes; PDNO).
  Explore potential biomarkers.
Assess the levels of the following biomarkers: 1,2-propanediol (PD) metabolites in serum | Change from baseline T0 (-15 minutes; placebo) to time point T6 (75 minutes; PDNO).
  Explore PD metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Kemi, PhD, Study Director — Attgeno AB
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Anaesthesiology and Intensive Care, Gothenburg
  - Örebro University Hospital, Vascular and Thoracic Department (Kärl-Thoraxkliniken), Örebro

IPD SHARING:
Plan to Share IPD: No